CLINICAL TRIAL: NCT06627829
Title: Effect of Different Grafting Material Following Surgically Facilitated Orthodontics Therapy: a Randomized Controlled Clinical Trial
Brief Title: Effect of Different Grafting Material Following Surgically Facilitated Orthodontics Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: American Academy of Periodontology Foundation (Unknown)
Responsible Party: Principal Investigator, Sahar Dowlatshahi, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-24-0478
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Malocclusion, Angle Class I
Keywords: orthodontic treatment
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group A (Experimental)
  Interventions: Device: Surgically facilitated orthodontics therapy (SFOT) using allograft
- Group B (Experimental)
  Interventions: Device: Surgically facilitated orthodontics therapy (SFOT) using xenograft
- Control group (Active Comparator)
  Interventions: Device: Usual care

INTERVENTIONS:
Device: Surgically facilitated orthodontics therapy (SFOT) using allograft — Participants will receive Surgically facilitated orthodontics therapy (SFOT) along with bone grafting using particulate allograft and collagen membrane, prior to orthodontics treatment.
  Arms: Group A
Device: Surgically facilitated orthodontics therapy (SFOT) using xenograft — Participants will receive SFOT using particulate xenograft and collagen membrane, prior to orthodontics treatment.
  Arms: Group B
Device: Usual care — Participants will have conventional orthodontics treatment with Invisalign aligners, without any surgical intervention
  Arms: Control group

SUMMARY:
The purpose of this study is to quantitatively investigate the radiographic changes of alveolar bone, and gingival tissue changes of the mandibular anterior teeth in experimental group A receiving SFOT using freeze-dried allograft with a collagen membrane, experimental group B receiving SFOT using particulate xenograft covered by a collagen membrane and control group receiving only orthodontics therapy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I/II
* Periodontal diagnosis of clinical gingival health or gingivitis on intact/reduced periodontium per 2017 American Academy of Periodontology (AAP) classification
* No history of periodontitis.
* Class I malocclusion
* Crowding of 4 mm or less on mandibular anterior incisors
* Incisor mandibular plane angle between 90-100 degrees
* No extractions indicated as part of the orthodontic treatment plan
* Keratinized tissue of at least 3mm

Exclusion Criteria:

* Patients who are current smokers
* Pregnancy
* Uncontrolled diabetes or other metabolic systemic conditions
* Presence of open bite or deep bite
* Spacing
* Excessive retroclined mandibular incisors
* Any contraindication to treatment or the material used if in the experimental groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2026-01-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
Change in horizontal bone thickness at the 3mm point from Cementoenamel junction (CEJ) (crestal level) on the mandibular incisors | from baseline to endpoint (Alignment visit, approximately 4 months after the start of orthodontics treatment)
Change in horizontal bone thickness at the 6mm point from CEJ (middle level) on the mandibular incisors | from baseline to endpoint (Alignment visit, approximately 4 months after the start of orthodontics treatment)
Change in horizontal bone thickness at the 9mm point from CEJ (apical level) on the mandibular incisors | from baseline to endpoint (Alignment visit, approximately 4 months after the start of orthodontics treatment)
Change in volume of three dimensional bone | from baseline to endpoint (Alignment visit, approximately 4 months after the start of orthodontics treatment)
Change in volume of three dimensional soft tissue | from baseline to endpoint (Alignment visit, approximately 4 months after the start of orthodontics treatment)

SECONDARY OUTCOMES:
Change in vertical bone level (VBL)from the CEJ | Baseline, at alignment (approximately 4 months after the start of orthodontics treatment).
Change in probing depth (PD) | Baseline, at alignment (approximately 4 months after the start of orthodontics treatment).
  PD is the distance from CEJ to base of gingival pocket
Change in clinical attachment level (CAL) | Baseline, at alignment (approximately 4 months after the start of orthodontics treatment).
  CAL is the distance between CEJ and base of the pocket
Change in width of keratinized tissue (WKT) at alignment | Baseline, at alignment (approximately 4 months after the start of orthodontics treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Dowlatshahi, DDS, MMSc, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No